CLINICAL TRIAL: NCT05640687
Title: The Study of Mesenchymal Stem Cells Treat Autoimmune Pulmonary Alveolar in Vitro
Brief Title: The Study of Mesenchymal Stem Cells Treat Autoimmune Pulmonary Alveolar Proteinosis in Vitro
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: 2020132
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Alveolar Proteinosis(PAP)
Keywords: aPAP; cell therapy; MSC
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aPAP
- healthy control

SUMMARY:
Autoimmune pulmonary alveolar proteinosis (aPAP) is a respiratory disease characterized by massive deposition of pulmonary surfactant in the alveoli, involving a variety of immune cells and factor disorders. However, there are certain limits in treatment at present. MSCs can improve the microenvironment in the alveoli by regulating immunity, thereby achieving a good therapeutic effect. The purpose of this study is to use the lavage fluid obtained after whole lung lavage with aPAP to isolate alveolar macrophages, and to use MSC to complete the verification of the efficacy of aPAP primary alveolar macrophages in vitro. A series of protocols including multi-factor detection, cell phenotype analysis and phagocytosis assay were used to evaluate the efficacy of MSCs on alveolar macrophages.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form before any research-related activities;
2. No gender restrictions, age ≥18 years old, and ≤75 years old;
3. Patients who need to receive whole lung lavage due to the needs of the disease, and the patient agrees to perform whole lung lavage. The standards are as follows:

   1. The diagnosis of aPAP is clear, and the anti-GM-CSF antibody in serum is greater than 5 μg/ml;
   2. PaO2 <65 mmHg;
   3. P(A-a)O2>40 mmHg;
   4. Intrapulmonary shunt >10%-12%.

Exclusion Criteria:

1. Suffering from multiple chronic respiratory diseases at the same time, including but not limited to chronic obstructive pulmonary disease, pulmonary fibrosis, and asthma;
2. Various malignant tumors or a history of malignant tumors;
3. Uncontrolled pulmonary or systemic infection;
4. Severe other systemic diseases: acute myocardial infarction, unstable angina pectoris, liver cirrhosis, acute glomerulonephritis, etc.;
5. Syphilis, HIV, HCV antibody positive;
6. Patients with coagulation disorders who cannot perform bronchoscopy, such as hemophilia, giant platelet syndrome, thrombocytopenia, etc.;
7. Severe renal impairment, serum creatinine > 1.5 times the upper limit of normal;
8. Liver disease or liver function damage: ALT, AST, total bilirubin > 2 times the upper limit of normal;
9. Have any coexisting medical conditions or diseases that the investigators judge may impair the development of this trial;
10. Social and mental disability, no legal capacity/limited capacity;
11. Refuse to sign the informed consent.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project recruited clinical patients who met the criteria for inclusion and exclusion from patients diagnosed with aPAP in the First Affiliated Hospital of Guangzhou Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-06 (Estimated)

PRIMARY OUTCOMES:
Genomics | 2022.12.31-2023.03.01

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China